CLINICAL TRIAL: NCT00867698
Title: A Phase 2, Multi-Center, Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Trial to Evaluate the Efficacy, Safety and Tolerability of AST-120 (Spherical Carbon Adsorbent) for 8 Weeks in the Treatment of Mild Hepatic Encephalopathy
Brief Title: AST-120 Used to Treat Mild Hepatic Encephalopathy
Acronym: ASTUTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ocera Therapeutics (Industry)
Responsible Party: Jeff Bornstein, MD, Ocera Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AST-MHE201
Record Dates: First submitted 2009-03-20; First posted 2009-03-24 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Mild Hepatic Encephalopathy
Keywords: Hepatic encephalopathy; Mild hepatic encephalopathy; HE; MHE; Cognitive impairment; Cognitive dysfunction; Liver Disease; Cirrhosis
MeSH Terms: conditions — Hepatic Encephalopathy; Cognitive Dysfunction; Liver Diseases; Fibrosis | interventions — AST 120

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AST-120 (6g) (Experimental): 2 grams TID
  Interventions: Drug: AST-120
- Placebo A (Placebo Comparator): 2 grams TID
  Interventions: Drug: AST-120
- AST-120 (12g) (Experimental): 4 grams TID
  Interventions: Drug: AST-120
- Placebo B (Placebo Comparator): 4 grams TID
  Interventions: Drug: AST-120

INTERVENTIONS:
Drug: AST-120 — AST-120
  Other Names: Spherical carbon adsorbent

SUMMARY:
The purpose of this study is to determine whether AST-120 is safe and effective in the treatment of mild hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed cirrhosis of any cause
2. Abnormal RBANS global summary score
3. Grade 0 or 1 hepatic encephalopathy by West-Haven Scale
4. MELD score < or = 25
5. Females must be postmenopausal, surgically incapable of bearing children or practicing a reliable method of birth control

Exclusion Criteria:

1. Previous participation in any trial involving AST-120
2. History of TIPS or surgically created portocaval shunt
3. Treatment for overt HE within the past 3 months
4. Use of lactulose, rifaximin, neomycin or other antibiotics in the past 7 days
5. Active alcohol abuse
6. Psychosis or organic brain syndromes due to alcohol or other causes
7. Use of interferon and sedating or cognition-altering drugs
8. Undergoing chemotherapy or radiotherapy for the treatment of cancer
9. Active GI bleeding within the past 3 months
10. Presence of an active infection
11. Presence of signs and symptoms of severe dehydration
12. Other major physical or major psychiatric illness within the past 6 months
13. Pregnant, breast feeding, or planning to become pregnant during the study
14. Using hormonal contraception as the only method of birth control

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Neurocognitive improvement, defined as the change in the global summary score of the RBANS at Week 8 compared to Baseline. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Bornstein, MD, Study Director — Ocera Therapeutics, Inc.
Locations (38):
- United States (38):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - UCSF - Fresno Community Regional Medical Center, Fresno, California
  - UCSD Medical Center, La Jolla, California
  - Scripps Clinic, San Diego, California
  - UCSD Medical Center, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida College of Medicine, Gainesville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami, Division of Hepatology / Center for Liver Disease, Miami, Florida
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - VA Medical Center / University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Delta Research Partners, LLC, Monroe, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconnes Medical Center, Harvard Medical School, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Weill Medical College of Cornell, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - New York Medical College, Valhalla, New York
  - University of Cincinatti, Cincinnati, Ohio
  - Case Western Reserve / MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Division of Hepatology, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of Southern Carolina, Charleston, South Carolina
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Advanced Liver Therapies, St. Luke's Episcopal Hospital/Baylor College of Medicine, Houston, Texas
  - Permian Research Foundation, Odessa, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - McGuire DVAMC, Richmond, Virginia